CLINICAL TRIAL: NCT02578030
Title: A Phase 1, Open-label Study of the Pharmacokinetics of d- and L-amphetamine After a Single Dose of SHP465 12.5 mg or 25 mg Administered to Children and Adolescents Aged 6 to17 Years With Attention-Deficit Hyperactivity Disorder (ADHD)
Brief Title: Pharmacokinetic Study in Children and Adolescents Aged 6 to 17 Years Who Have Been Diagnosed With ADHD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHP465-111
Record Dates: First submitted 2015-10-05; First posted 2015-10-16 (Estimated); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SHP465 12.5 mg (Experimental): A single dose of SHP465 12.5 mg for Subjects aged 6-12 years
  Interventions: Drug: SHP465 12.5mg
- SHP465 25 mg (Experimental): A single dose of SHP465 25 mg for Subjects aged 13-17 years
  Interventions: Drug: SHP465 25mg

INTERVENTIONS:
Drug: SHP465 12.5mg
  Arms: SHP465 12.5 mg
Drug: SHP465 25mg
  Arms: SHP465 25 mg

SUMMARY:
To provide additional, required information on the pharmacokinetic profile of SHP465 in the targeted population (children and adolescents aged 6-17 years of age with ADHD).

ELIGIBILITY:
Inclusion Criteria:

1. Age 6 to 17 years inclusive at the time of consent/assent. The date of signature of the informed consent/assent is defined as the beginning of the Screening Period. This inclusion criterion will only be assessed at the first screening visit.
2. Male, or non-pregnant, non-lactating female who agrees to comply with any applicable contraceptive requirements of the protocol or females of non-childbearing potential.
3. Subject meets Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) criteria for a primary diagnosis of ADHD based on an accepted ADHD diagnostic instrument and documented in the subject's medical record. Subject's ADHD is currently adequately controlled with an amphetamine-based product.
4. Subject is functioning at an age appropriate level intellectually, as determined by the investigator.
5. Must be considered "healthy". Healthy status is defined by absence of evidence of any active or chronic disease other than their ADHD following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead ECG, hematology, blood chemistry, and urinalysis.
6. Ability to swallow a capsule of investigational product whole.

Exclusion Criteria:

1. Current use of any ADHD medication other than an amphetamine-based product.
2. History of any hematological, hepatic, respiratory, cardiovascular, renal, neurological or psychiatric disease, gall bladder removal, or current or recurrent disease other than their ADHD
3. Current or relevant history of physical or psychiatric illness, any medical disorder that may require treatment
4. Subject has a current, controlled or uncontrolled, comorbid psychiatric diagnosis with significant symptoms
5. Subject meets DSM-V diagnosis of conduct disorder.
6. Subject is considered a suicide risk in the opinion of the investigator, has previously made a suicide attempt, or is currently demonstrating active suicidal ideation.
7. Subject is underweight based on Centers for Disease Control and Prevention (CDC) body mass index (BMI)- for-age sex-specific values
8. Subject is significantly overweight based on CDC BMI-for-age sex specific values
9. Subject has a known history of symptomatic cardiovascular disease, advanced arteriosclerosis, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, coronary artery disease, or other serious cardiac problems
10. Subject has a concurrent chronic or acute illness, disability, or other condition that might confound the results of safety assessments conducted in the study
11. Subject has a history of seizure, a chronic or current tic disorder, or a current diagnosis of Tourette's Disorder. Subject has a history of tics that are judged to be exclusionary.
12. Subject's blood pressure measurements exceed the 90th percentile for age, sex, and height
13. Subject has a known history of hypertension.
14. Subject has a known family history of sudden cardiac death or ventricular arrhythmia.
15. Subject has any clinically significant ECG or clinically significant laboratory abnormality
16. Subject has abnormal thyroid function
17. Known or suspected intolerance or hypersensitivity to the investigational product(s), closely-related compounds, or any ingredients.
18. History of alcohol or other substance abuse within the last year. Subjects with a lifetime history of amphetamine, cocaine, or other stimulant abuse and/or dependence will be excluded.
19. Use Within 30 days prior to the first dose of investigational product:

    * have used an investigational product
    * have been enrolled in a clinical study (including vaccine)
    * have had any substantial changes in eating habits
20. A positive screen for alcohol or drugs of abuse. A positive hepatitis B surface antigen (HBsAg); hepatitis C virus (HCV); or HIV antibody screen.
21. Use of tobacco in any form in the last 30 days
22. Prior screen failure, enrollment, or participation in this study.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2015-10-24 (Actual); Primary Completion 2015-11-10 (Actual); Study Completion 2015-11-10 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Drug Concentration (Cmax) of Dextroamphetamine (d-amphetamine) in Plasma | Pre-dose, 2, 4, 6, 8, 10, 12, 24, 48, 72 hours post-dose
  Maximum concentration occurring at time of maximum observed concentration of d-amphetamine during a dosing interval.
Maximum Observed Drug Concentration (Cmax) for Levoamphetamine (l-amphetamine) in Plasma | Pre-dose, 2, 4, 6, 8, 10, 12, 24, 48, 72 hours post-dose
  Maximum observed concentration of l-amphetamine during a dosing interval.
Time to Reach Maximum Observed Drug Concentration (Tmax) of Dextroamphetamine (d-amphetamine) in Plasma | Pre-dose, 2, 4, 6, 8, 10, 12, 24, 48, 72 hours post-dose
  Time to reach maximum observed drug concentration of d-amphetamine during a dosing interval.
Time to Reach Maximum Observed Drug Concentration (Tmax) of Levoamphetamine (l-amphetamine) in Plasma | Pre-dose, 2, 4, 6, 8, 10, 12, 24, 48, 72 hours post-dose
  Time to reach maximum observed drug concentration of l-amphetamine during a dosing interval.
Area Under the Curve From Zero to Infinity (AUC0-infinity) of Dextroamphetamine (d-amphetamine) in Plasma | Pre-dose, 2, 4, 6, 8, 10, 12, 24, 48, 72 hours post-dose
  AUC0-infinity was calculated using the observed value of the last non-zero concentration of d-amphetamine in plasma.
Area Under the Curve From Zero to Infinity (AUC0-infinity) of Levoamphetamine (l-amphetamine) in Plasma | Pre-dose, 2, 4, 6, 8, 10, 12, 24, 48, 72 hours post-dose
  AUC0-infinity was calculated using the observed value of the last non-zero concentration of l-amphetamine in plasma.
Area Under the Curve From Zero to Last Measurable Concentration (AUClast) of Dextroamphetamine (d-amphetamine) in Plasma | Pre-dose, 2, 4, 6, 8, 10, 12, 24, 48, 72 hours post-dose
  Area under the curve from the time of dosing to the last measurable concentration of d-amphetamine in plasma.
Area Under the Curve From Zero to Last Measurable Concentration (AUClast) of Levoamphetamine (l-amphetamine) in Plasma | Pre-dose, 2, 4, 6, 8, 10, 12, 24, 48, 72 hours post-dose
  Area under the curve from the time of dosing to the last measurable concentration of l-amphetamine in plasma.
Terminal Half-life (t½) of Dextramphetamine (d-amphetamine) in Plasma | Pre-dose, 2, 4, 6, 8, 10, 12, 24, 48, 72 hours post-dose
  Terminal half-life is the time measured for the plasma concentration of d-amphetamine to decrease by one half.
Terminal Half-life (t½) of Levoamphetamine (l-amphetamine) in Plasma | Pre-dose, 2, 4, 6, 8, 10, 12, 24, 48, 72 hours post-dose
  Terminal half-life is the time measured for the plasma concentration of l-amphetamine to decrease by one half.
Total Body Clearance for Extravascular Administration (CL/F) of Dextroamphetamine (d-amphetamine) | Pre-dose, 2, 4, 6, 8, 10, 12, 24, 48, 72 hours post-dose
  Total body clearance for extravascular administration of d-amphetamine divided by the fraction of dose absorbed.
Total Body Clearance for Extravascular Administration (CL/F) of Levoamphetamine (l-amphetamine) | Pre-dose, 2, 4, 6, 8, 10, 12, 24, 48, 72 hours post-dose
  Total body clearance for extravascular administration of l-amphetamine divided by the fraction of dose absorbed.
Volume of Distribution After Extravascular Administration (Vz/F) of Dextroamphetamine (d-amphetamine) | Pre-dose, 2, 4, 6, 8, 10, 12, 24, 48, 72 hours post-dose
  Volume of distribution for d-amphetamine based on the terminal phase following extravascular administration divided by the fraction of dose absorbed.
Volume of Distribution After Extravascular Administration (Vz/F) of Levoamphetamine (l-amphetamine) | Pre-dose, 2, 4, 6, 8, 10, 12, 24, 48, 72 hours post-dose
  Volume of distribution for l-amphetamine based on the terminal phase following extravascular administration divided by the fraction of dose absorbed.

SECONDARY OUTCOMES:
Participants with Treatment-emergent Adverse Events (TEAEs) | From start of study drug administration up to follow-up (up to 9 days)
  An adverse event (AE) was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. An AE was considered as treatment-emergent (TEAE) if it had a start date and time on or after the dose of investigational product and no later than 72 hours after dosing, or if it had a start date and time before the date and time of the dose of investigational product, but increased in severity on or after the date and time of the dose of investigational product and no later than 72 hours after dosing.
Number of Participants With TEAE Related to Vital signs, Electrocardiogram (ECG), and Clinical Laboratory Tests | From start of study drug administration up to follow-up (up to 9 days)
  An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Vital signs included blood pressure, pulse rate, respiratory rate, and body temperature. ECG was analysed as 12-lead ECG. Clinical laboratory test is considered for biochemistry, Hematology and Urinalysis.
Number of Participants With Suicidal Behavior and / or Ideation ("Yes" Response) on the Columbia Suicide Severity Rating Scale (C-SSRS) | Baseline up to Day 4
  C-SSRS is a clinician rated assessment of suicidal behavior and / or intent categorized as: Suicidal behavior=a "yes" response to any of 5 suicidal behavior questions (preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide); Suicidal ideation=a "yes" response to any one of 5 suicidal ideation questions which includes wish to be dead, and 4 different categories of active suicidal ideation (thought, thought with method, thought with intent, thought with plan and intent).

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (3):
- United States (3):
  - QPS MRA, Miami, Florida
  - Center for Psychiatry and Behavioral Medicine, Inc., Las Vegas, Nevada
  - Houston Clinical Research, Houston, Texas